CLINICAL TRIAL: NCT02763176
Title: Measuring hCG Levels in Pregnant Women: a Prenatal Study of hCG Using MLPT and Serum Testing
Brief Title: Measuring hCG Levels in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 6007
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: hCG
Keywords: hCG testing, multi-level pregnancy test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine for hCG measurement
Oversight: Data Monitoring Committee: No

SUMMARY:
This study seeks to assess trends in hCG between the 9th and 12th weeks of gestation. Women presenting at prenatal care at the study site who are 70 days gestation or less will be offered participation in the study. 75 consenting women will be asked to provide urine for an MLPT and to have blood drawn for hCG serum testing at 56-63 days, 64-70 days, and 71-77 days' gestation, and 75 consenting women will be asked to provide urine for an MLPT and to have blood drawn for hCG serum testing at 64-70 days, 71-77 days, and 78-84 days' gestation.

DETAILED DESCRIPTION:
Women presenting at the study site for a prenatal visit, and who are ≤ 70 days' gestation, will be offered participation in the study. Efforts will also be made to recruit patients through physician or treating health care professional referral and advertisements. One hundred and fifty consenting women will be enrolled. Up to three additional study visits will be scheduled: At the enrollment, if an ultrasound-confirmed gestational age is not available in the woman's medical record, a transvaginal ultrasound will be performed. If the woman is 56-63 days gestation on the day of enrollment, she will be asked to return weekly until she reaches 71-77 days. If the woman is 64-70 days gestation, she will be asked to return weekly until she reaches 78-84 days. If the woman is less than 56 days gestation, she will be asked to return for the three research visits at the appropriate time to provide the urine samples and blood draws. Women will have one visit during each of their three assigned gestational age weeks. At each visit, women will provide a urine sample for an MLPT and have a blood draw to measure serum hCG.

ELIGIBILITY:
Inclusion Criteria:

* Intrauterine pregnancy <= 70 days' gestation
* Be in general good health
* English speaking competency
* Be willing and able to sign consent forms
* Agree to comply with the study procedures, including returning for three study visits that each involve a blood draw and urine pregnancy test for measuring hCG

Exclusion Criteria:

* Women less than 18 years of age.
* Any women not meeting the inclusion criteria listed above will be excluded from participating in the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women seeking prenatal care.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
hCG trends | Between 56-84 days gestation
  To ascertain the proportion of women with decreases in hCG between 56-84 days gestation

IPD SHARING:
Plan to Share IPD: No